CLINICAL TRIAL: NCT07030010
Title: Examining the Efficacy of a Commercially Available Multi-ingredient Liquid Tonic Drink on Postprandial Glycemia in Men and Women With Overweight and/or Obesity.
Brief Title: Effect of a Liquid Tonic Drink on Post-meal Glucose and Insulin Responses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Australian Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2025-4309HC
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Overweight or Obese Adults
Keywords: Postprandial hormones; Mixed meal challenge; Tonic drink
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: Two arm, cross-over design where all participants will receive both conditions in different orders
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All researchers involved in undertaking the study and analysing the data will be blinded. Participants will be blinded. The dietitian preparing and serving the meal and drink will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tonic drink (Active Comparator): This arm will receive the tonic drink on their first postprandial challenge
  Interventions: Other: Breakfast meal challenge with tonic drink
- Placebo drink (Placebo Comparator): This arm will receive the placebo drink on their first postprandial challenge
  Interventions: Other: Breakfast meal challenge with placebo drink

INTERVENTIONS:
Other: Breakfast meal challenge with tonic drink — High-carbohydrate containing breakfast meal with the addition of the tonic drink
  Arms: Tonic drink
Other: Breakfast meal challenge with placebo drink — High-carbohydrate containing breakfast meal with the addition of the placebo drink
  Arms: Placebo drink

SUMMARY:
A randomised, double blinded, placebo-controlled crossover design clinical trial conducted at the Mary MacKillop Institute for Health Research (MMIHR, Australian Catholic University) for individuals with overweight/ obesity. This study will measure the postprandial glucose and hormone responses to a high-carbohydrate meal with/ without a liquid tonic drink.

DETAILED DESCRIPTION:
Twenty individuals living with overweight/ obesity will be invited to attend the university laboratories on 2 separate occasions to participate in a postprandial (meal) challenge. Participants will consume the same high-carbohydrate meal on each visit, with or without a liquid tonic drink. This will be a cross-over design study, where participants will consume a placebo drink on the alternate visit. Participants will remain in the laboratory for 3-hours following the meal with a venous cannula in place, and have blood samples taken at regular timepoints. Blood samples will be analysed for glucose and appetite hormones. Participants will also wear a continuous glucose monitor throughout the period which encapsulates both study trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥30-64 years
* Body Mass Index (BMI) of ≥27.0 kg/m2

Exclusion Criteria:

* younger than 30 or 65 years or older,
* a BMI less than 27.0 kg/m2,
* have an allergy to any of the components in the plant-based tonic (see section 6),
* pregnant or breastfeeding,
* regularly skipping breakfast (i.e. not consuming breakfast on 5/7 days per week),
* any diagnosed metabolic (e.g. diabetes), endocrine (e.g. hyperthyroidism), gastrointestinal (e.g. Crohn's) or cardiovascular (e.g. heart failure) abnormalities,
* on an energy-restricted diet; significant weight fluctuation in the previous 3 months (>5% body weight),
* high alcohol consumption (>14 units/week) (as per Alcohol Drink Guidelines),
* medication that is used to treat blood glucose,
* unable to attend in person testing sessions, or
* unable or unwilling to provide blood samples.

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
3-hour postprandial glucose incremental area under the curve | 3 hours
  Venous glucose concentrations measured over the 3 hour period following consumption of the breakfast meal and tonic drink/ placebo, and calculated using the trapezoid method, with T0 concentration as baseline

SECONDARY OUTCOMES:
3-hour postprandial insulin incremental area under the curve | 3-hours
  Venous insulin concentrations measured over the 3 hour period following consumption of the breakfast meal and tonic drink/ placebo, and calculated using the trapezoid method, with T0 concentration as baseline
3-hour interstitial postprandial glucose incremental area under the curve | 3 hours
  The interstitial glucose levels observed for the 3 hours following consumption of the breakfast meal and tonic drink/placebo using continuous glucose monitors
Matsuda index (Marker of whole-body postprandial insulin sensitivity) | 3 hours
  This marker takes into account the 3- hour postprandial venous blood glucose and insulin measurements observed
Venous blood C-peptide responses | 3 hours
  3-hour postprandial C-peptide responses measured in venous blood as a marker of insulin secretion
Venous blood insulin to glucagon ratio's at baseline (T0) and 30 minutes (T30) | 30 minutes
  Ratio of venous blood insulin to glucagon at baseline and 30 minutes (T0, T30) as a marker of hepatic glucose production.

CONTACTS AND LOCATIONS:
Overall Officials: Leonidas Karagounis, PhD, Principal Investigator — Australian Catholic University
Locations (1):
- Australian Catholic University, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the corresponding author for a period of 36 months from publication, upon reasonable request for academic use. The data will not be made publicly available, as it contains information that could compromise research participant consent.
Supporting Information: Study Protocol
Access Criteria: Reasonable requests of data for academic use will be considered. Requests can be made to the corresponding author of the publication. Data will not be made publicly available as it contains information that could compromise research participant consent.